CLINICAL TRIAL: NCT04728269
Title: Exploratory Study to Assess the Impact of a Cosmetic Product (Lactibiane Topic AD) on Skin Flora and Skin Reinforcement Barrier in Mild to Moderate Atopic Dermatitis
Brief Title: Exploratory Study on Lactibiane Topic AD on Skin Flora and Barrier Reinforcement in Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DEABIOM
Record Dates: First submitted 2021-01-14; First posted 2021-01-28 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactibiane topic AD (Experimental): Cosmetical product Lactibiane Topic AD
  Interventions: Other: Lactibiane Topic AD
- Placebo (Placebo Comparator): Placebo made with the same base as the cosmetical product
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Lactibiane Topic AD — Application of Lactibiane topic AD twice a day (morning and evening) on one lesional area
  Arms: Lactibiane topic AD
Other: Placebo — Application of placebo twice a day (morning and evening) on the symmetrical lesional area
  Arms: Placebo

SUMMARY:
This exploratory study aims to evaluate the impact of a cosmetic product (Lactibiane Topic AD) vs placebo on skin flora and skin reinforcement barrier in mild to moderate atopic dermatitis using biometrological, biological and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with mild to moderate AD defined as SCORAD≤40 (Eichenfield et al. JAAD 2014).
* Subject with at least two symmetric AD lesions with comparable severity: Located either on upper extremities (left and right arms except hands) or lower extremities (left and right legs except feet), With an erythema ≥ 1 (mild to severe intensity), With a lesional area score ≥ 4 on both lesions with an authorized delta of two points between the two lesions, With a sufficient extent to allow all the investigations.
* Subject with I, II, III or IV skin phototype (according to Fitzpatrick's scale).
* For woman of childbearing potential (defined as all women physiologically capable of becoming pregnant): Negative urine pregnancy test at inclusion visit. Use of a highly effective method of birth control* during the study. * A highly effective method of birth control is defined as one which results in a low failure rate (less than 1%) when used consistently and correctly, such as implants, combined oral contraceptives, intrauterine device, double barrier methods (e.g. condom with spermicide), sexual abstinence or vasectomized partner.
* Subject with health insurance coverage according to local regulation.
* Subject having given his written informed consent.

Exclusion Criteria:

* Subject having a known hypersensitivity, allergy or contraindication to any ingredients contained within the investigational product or placebo.
* Subject having exposed his skin to natural or artificial UV within 8 weeks prior to the inclusion visit or intending to expose his skin during the study.
* Subject having performed phototherapy within 8 weeks prior to the inclusion visit or intending to perform phototherapy during the study.
* Subject having performed another physical treatment (e.g radiotherapy…) on the investigational areas within 6 months prior to the inclusion visit or intending to perform it during the study.
* Subject treated with systemic non-steroidal anti-inflammatory drugs (≥3 days) within 1 week before the inclusion visit.
* Subject treated with biological immunosuppressive drugs within 12 weeks prior to the inclusion visit or intending to be treated with it during the study.
* Subject treated with non-biological immunosuppressive drugs within 4 weeks prior to the inclusion visit or intending to be treated with it during the study.
* Subject treated with systemic corticoids within 1 week prior to the inclusion visit or planed during the study.
* Subject treated with systemic antibiotics within 7 days prior to the inclusion visit or planed during the study.
* Subject having applied topical immunomodulators, non-steroidal anti-inflammatory, corticoids or antihistamines on investigational limbs within 1 weeks prior to the inclusion visit.
* Subject having applied topical antibiotics or disinfectants on investigational limbs within 2 weeks prior to the inclusion visit.
* Subject having applied any other topical and/or care product after the last grooming prior to the inclusion visit.
* Subject having applied water or care product (except hands cleaning) within 12 hours prior to the inclusion visit.
* Subject having started, modified or stopped any other treatment/product within 4 weeks prior to the inclusion visit or intending to do so during the study that according to the investigator's judgment, could interfere with study results.
* Subject having significant medical condition that according to the investigator's judgment, deems inappropriate for study participation (e.g present or past malignancy, present or past skin condition…).
* Subject having significant dermatological condition or sign (e.g disease, scare, abundant hairiness, tanning mark…) that according to the investigator's judgment, could limit the observations or/and interfere with the interpretations.
* Subject taking part or having participated in another clinical study within 2 weeks prior to the inclusion visit.
* Subject under legal guardianship or incapacitation.
* Subject linguistically or psychologically unable of signing informed consent form and unable to comply with the protocol requirements according to the investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Change in skin flora composition | from baseline (Day 0) at Day 21
  16S rRNA sequencing, qPCR
Change in skin flora composition | from baseline (Day 0) at Day 14
  16S rRNA sequencing, qPCR

SECONDARY OUTCOMES:
Skin barrier status | Day 0, Day 14, Day 21
  TransEpidermal Water Loss (TEWL)
Patient Oriented SCORing Atopic Dermatitis | Day 0, Day 14, Day 21
  Patient Oriented SCORing Atopic Dermatitis (POSCORAD): 0 - 103 (Higher values represent a worse outcome)
SCORing Atopic Dermatitis | Day 0, Day 14, Day 21
  SCORing Atopic Dermatitis (SCORAD) : 0 - 103 (Higher values represent a worse outcome)
Clinical severity of lesional areas | Day 0, Day 14, Day 21
  Scoring of lesional area by subject and investigator : 0-18 (Higher values represent a worse outcome)
Manifestation of adverse local reactions | From Day 0 to Day 21
  Subjects will use a diary to document any potential adverse reactions observed after product application

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de Recherche Clinique en Immunologie - Lyon Sud, Pierre-Bénite, France